CLINICAL TRIAL: NCT07351734
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetic Characteristics of JKN2403 Tablets in Patients With Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Trial of JKN2403 in COPD
Acronym: COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joincare Pharmaceutical Group Industry Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKN2403-IIa; JKN2403-IIa (Other Grant/Funding Number: Joincare Pharmaceutical Group Industry Co., Ltd)
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dose1 of JKN2403 Tablets, once daily orally (Experimental): dose1 of JKN2403 Tablets once daily orally, for 24 weeks
  Interventions: Drug: JKN2403 Tablets
- dose2 of JKN2403 Tablets once daily orally (Experimental): dose2 of JKN2403 Tablets once daily orally, for 24 weeks
  Interventions: Drug: JKN2403 Tablets
- dose3 of JKN2403 Tablets once daily (Experimental): dose3 of JKN2403 Tablets once daily orally, for 24 weeks
  Interventions: Drug: JKN2403 Tablets
- Placebo once daily (Placebo Comparator): Placebo once daily orally, for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JKN2403 Tablets — JKN2403 Tablets once daily orally, for 24 weeks
  Arms: dose1 of JKN2403 Tablets, once daily orally; dose2 of JKN2403 Tablets once daily orally; dose3 of JKN2403 Tablets once daily
Drug: Placebo — Placebo
  Arms: Placebo once daily

SUMMARY:
The goal of this clinical trial is to learn if drug JKN2403 works to treat moderate-to-severe COPD in adults. It will also learn about the safety and pharmacokinetic characteristics of drug JKN2403. The main questions it aims to answer are:

Does drug JKN2403 reduce the incidence of AECOPD or improve the quality of life or alleviate symptoms related to COPD?

Researchers will compare drug JKN2403 to a placebo (a look-alike substance that contains no drug) to see if drug JKN2403 works to treat moderate-to-severe COPD.

Participants will:

Take drug JKN2403 or a placebo every day for 24 weeks Visit the clinic once every four weeks for checkups and tests Keep a diary of their symptoms and the number of times they use a rescue inhaler

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent; able and willing to comply with study procedures.
* Adults with documented COPD diagnosis and medical history consistent with guideline criteria.
* Relevant exposure history consistent with COPD (e.g., smoking).
* On stable, guideline-based maintenance COPD therapy prior to randomization, per investigator judgment.
* Protocol-defined exacerbation history, symptom burden, and lung function at screening.

Exclusion Criteria:

* Current or past asthma, or other clinically significant respiratory disease that may confound assessment.
* Clinically significant uncontrolled comorbidities that increase risk or interfere with participation/outcomes.
* Immunodeficiency/immune dysregulation, active autoimmune disease requiring systemic immunosuppression, or significant opportunistic infection history.
* Active clinically significant infection or recent infection requiring systemic therapy; recent protocol-defined COPD exacerbation.
* Current/recent malignancy (except low-risk, adequately treated cancers per protocol) or clinically significant abnormal screening labs.
* Prohibited recent vaccines or therapies, prior relevant biologic/targeted therapy exposure, severe hypersensitivity to biologics/IMP, - pregnancy/breastfeeding, or inability to comply (including substance abuse), per investigator judgment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The annualized incidence rate of moderate to severe AECOPD | at 24 months
The duration from the first administration to the first occurrence of moderate to severe AECOPD | at 24 months

SECONDARY OUTCOMES:
trough (pre-bronchodilator) FEV1 | at 4, 8, 12 ,16, 20 and 24 weeks
quality of life（SGRQ score） | at 4, 8,12, 16, 20 and 24 weeks
quality of life (CAT score) | at 4, 8,12, 16, 20 and 24 months
The annualized incidence rate of CID | at 24 weeks
The duration from the first administration to the first occurrence of CID | at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No